CLINICAL TRIAL: NCT05865223
Title: Title Comparison Of Mackenzie Exercise Program Versus Routine Physical Therapy Management On Pain , Range Of Motion And Function in Patient With Chronic Mechanical Neck Pain
Brief Title: Comparison Of Mackenzie Exercise Program Versus Routine Physical Therapy Management in Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/RCR&AHS/23/0018
Record Dates: First submitted 2023-04-18; First posted 2023-05-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mckenzie exercise program (Experimental): Group A Week 0 : Hot pack for 15 minutes, mackenzie extension exercise program for cervical regions and mobilization with movement at cervical regions for improving flexion, extension, side flexion and rotation. 3 sets of painless glides of 10 repetitions were given, with 1 minute rest between sets.
  * Week 2 & 4: Hot pack for 15 minutes, mckenzie exercise program at cervical region with the progression in repetition and MWM at cervical regions and then we will add progression.5 sets of painless glides of 10 repetitions were given, with 3 minute rest between sets.
  * Week 3 & 6: Hot pack for 15 minutes, mckenzie exercise program for cervical region and MWM at cervical region . 5 sets of painless glides for 10 repetitions were given. Progression can be introduced by increasing number of repetitions performed exercises for 3 weeks.
  Interventions: Other: Mckenzie exercise program
- conventional physical therapy (Active Comparator): A routine physical therapy(joint mobilization,hot pack and home exercise program) treatment and hot pack for 15 minutes.
  Interventions: Other: Conventional Physical therapy

INTERVENTIONS:
Other: Mckenzie exercise program — MacKenzie extension exercise program for cervical spine
  Arms: Mckenzie exercise program
Other: Conventional Physical therapy — hot pack for 15 minutes will be given followed by joint mobilization,and home exercise program.
  Arms: conventional physical therapy

SUMMARY:
Study will be a Randomized clinical trial to check comparison of mckenzie exercise program versus routine physical therapy management on pain, range of motion and function in patients with chronic neck pain so that we can devise a treatment protocol.Total fifty subjects will be included in this study .Out of total 25 will be randomly allocated via lottery method in group 1 and 25 will be allocated in group 2. Group 1 will receive mckenzie exercise program and routine physical therapy(Joint mobilization, hot pack for 15 minutes and home exercise program) while Group 2 will receive only routine physical therapy (Joint mobilization , hot pack for 15 min and home exercise program). All patients will be treated for 12 sessions, two sessions per week for 6 weeks. Neck pain and disability index consist of two parts, part one which assesses pain severity and part two which assesses functional disability. Study setting will be services hospital. Assesment will be done at 0 week, 4week, 8week and 12weeks. Data was analysed by using SPSS version 26.

DETAILED DESCRIPTION:
Neck pain is a key public health issue that affects the human beings with reduction productivity and quality of life and produced significant socioeconomic burden on society.The purpose of this study to determine the effectiveness of Mckenzie exercise program and routine physical therapy management on pain range of motion and function in patient with chronic mechanical neck pain. Patients of both gender, neck pain for at least 3 months and age 25-55 years will be included. Patients having history of trauma, vertebral fracture, congenital disorder, ankylosing spondylitis, tumour, pott's disease and any bony or soft tissue systematic disease will be excluded. The main objective of this study is to evaluate pain level and effect of Mackenzie protocol for individuals suffering from chronic neck pain.

The tools used will be Neck disability index score (NDI), Numeric Pain Rating Scale (NPRS) and Goniometer for outcome measure pain, range of motion and function. Study will be conducted into 2 groups, each group will have 12 patients and comparisons of two groups will be evaluated. One group will receive Mckenzie exercise program and Routine physical therapy (Joint Mobilization, Hot pack and home exercise program) for 12 weeks and 2 days a week for 40 min each session and other group will receive Routine physical therapy (Joint mobilization, Hot pack and home exercise plan) for 12 weeks and 2 days a week for 30 min each session. Assessment will be done at 0 weeks, 4 week, 8 week and 12 week.Both groups received hot packs for 15 minutes for warming up.

ELIGIBILITY:
Inclusion Criteria:

* Both Gender
* Neck pain for at least 3 months
* Age 25-55 years old

Exclusion Criteria:

* • History of trauma

  * Vertebral Fracture
  * Congenital disorder
  * Ankylosing spondylitis
  * Tumour
  * Pott's Spine
  * Any bony or soft tissue systemic disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | up to 12 weeks
  Patients are asked to circle the number on a Numerical Rating Scale (NRS) that best describes their level of discomfort between 0 and 10, 0 and 20, or 0 and 100. The lower limit often denotes "the least amount of suffering ," whereas zero typically denotes "no pain at all."
Universal Goniometer for range of motion measurement | up to 12 weeks
  The most popular and reliable approach for determining shoulder range of motion (ROM) is by utilizing a goniometer. A goniometer is a straightforward instrument that has two arms joined at a hinge. The goniometer's second arm would be used to measure the joint angle while the physiotherapist placed one arm of the patient against the patient's body
Neck disability index (NDI) | up to 12 weeks
  The Neck Disability Index (modification of the oswestry low back pain disability index) scale scores range from 0 to 5 and the total score is the sum of the item scores possible range 0 no pain to 100 maximal pain

CONTACTS AND LOCATIONS:
Overall Officials: Zanam Nasir, MS*, Principal Investigator — Riphah International University
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Aziem AA, Mohamed RR, Draz AH, Azab AR, Hegazy FA, Diab RH. The effect of McKenzie protocol vs. deep neck flexor and scapulothoracic exercises in subjects with chronic neck pain - a randomized controlled study. Eur Rev Med Pharmacol Sci. 2022 May;26(9):3138-3150. doi: 10.26355/eurrev_202205_28731. PMID 35587064
- [Background] Guez M, Hildingsson C, Nilsson M, Toolanen G. The prevalence of neck pain: a population-based study from northern Sweden. Acta Orthop Scand. 2002 Aug;73(4):455-9. doi: 10.1080/00016470216329. PMID 12358121
- [Background] Farooq MN, Mohseni-Bandpei MA, Gilani SA, Ashfaq M, Mahmood Q. The effects of neck mobilization in patients with chronic neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2018 Jan;22(1):24-31. doi: 10.1016/j.jbmt.2017.03.007. Epub 2017 Mar 4. PMID 29332752
- [Background] Letafatkar A, Rabiei P, Alamooti G, Bertozzi L, Farivar N, Afshari M. Effect of therapeutic exercise routine on pain, disability, posture, and health status in dentists with chronic neck pain: a randomized controlled trial. Int Arch Occup Environ Health. 2020 Apr;93(3):281-290. doi: 10.1007/s00420-019-01480-x. Epub 2019 Oct 25. PMID 31654125
- [Background] Swenson RS. Therapeutic modalities in the management of nonspecific neck pain. Phys Med Rehabil Clin N Am. 2003 Aug;14(3):605-27. doi: 10.1016/s1047-9651(03)00038-x. PMID 12948344
- [Background] Kjellman G, Oberg B. A randomized clinical trial comparing general exercise, McKenzie treatment and a control group in patients with neck pain. J Rehabil Med. 2002 Jul;34(4):183-90. doi: 10.1080/16501970213233. PMID 12201614